CLINICAL TRIAL: NCT05499988
Title: The Importance of Blastocyst Diamater and Its Correlation to Reproductive Outcomes in PGT-A Cases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ganin Fertility Center (Other)
Responsible Party: Principal Investigator, Eman Hasanen, Embryologist, Ganin Fertility Center
Other Study IDs: GFC-006
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Infertility
Keywords: Blastocyst diameter; PGT-A; Time lapse; Blastocyst survival; TE biopsy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Trophoectoderm samples were taken from day 5 or 6 blastocysts for PGT-A
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Morphometric measurement of blastocyst diameter was taken on the day of trophoectoderm biopsy. PGT-A was done using NGS platform, followed by thawing and transfer of euploid blastocyts. Follow up of the Pregnancy and implantation rates is done and recorded to study the correlation between the diameter and reproductive outcomes of the blastocyst.

DETAILED DESCRIPTION:
Blastocyst morphological grading proposed by Gardner and Schoolcraft including the expansion degree, inner cell mass, and trophoectoderm assessment has proved its importance. Blastocyst expansion degree that can presented in diameter is linked to the blastocyst implantation and overall success.

In order to evaluate the importance of blastocyst diameter in PGT-A cases, measurements will be taken on the day of trophoectoderm biopsy TE (diameter in μm), followed by TE biopsy using flicking technique. Next, PGT-A will be done using NGS platform and results will be confirmed using PGT-ai. Thawing of euploid blastocyst will take place and expansion degree, survival rate will be recorded. Patient will be followed up for the clinical pregnancy and implantation rates.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-45 years old
* Male aged 18-60 years old
* ICSI cases having PGT-A for their blastocysts
* Must have their blastocysts cultured in time lapse incubator

Exclusion Criteria:

* Presence of any of the endometrial factors that affect embryo implantation such as hydrosalpings, adenomyosis or previous uterine infection
* Any contradictions to undergoing in vitro fertilization or gonadotropin stimulation
* Use of donor oocytes or sperm
* Use of gestational carrier

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ICSI cases that have planned to do PGT-A for their blastocysts, oocytes were cultured in time lapse incubators from day 0-6. Female aged between 18 and 45 years old can be included. PGT-A was done using next generation sequencing (NGS) platform and their results were confirmed using PGT-ai.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Blastocoele re-expansion degree | Two hours post thawing
  Defined as the degree of blastocoele re-expansion and presented in %
Pregnancy rate | 15 days post embryo transfer
  Defined as clinical pregnancy per transfer
Implantation rate | 6-8 weeks of pregnancy
  Defined as number of gestational sacs with fetal heart beat, shown by ultrasound in gestational week 6 over number of embryo transferred.
Blastocyst survival rate | Two hours post thawing
  Defined as the proportion of blastocysts that showed expansion degree ≥50% and their cells remained intact after thawing and re-expansion

CONTACTS AND LOCATIONS:
Overall Officials: Eman Hasanen, BSc., Principal Investigator — Ganin Fertility Center; Manar Hozayen, MSc., Principal Investigator — Ganin Fertility Center; Amr Elshimy, BSc., Principal Investigator — Ganin Fertility Center; Hanaa Alkhader, Principal Investigator — Ganin Fertility Center; Hosam Zaki, MSc, FRCOG, Study Director — Ganin Fertility Center; Samar Gamal, BP, Principal Investigator — Ganin Fertility Center
Locations (1):
- Ganin Fertility Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP